CLINICAL TRIAL: NCT07319858
Title: The Effect of Using Multifunctional Baby Carrier on Physiological Parameters, Pain and Sleep Status in Babies With Heart Surgery
Brief Title: The Effect of Using Multifunctional Baby Carrier With Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aynur Baykal, PHD STUDENT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IUC-PHD-NURS-2025-01
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Surgery
Keywords: nursing; pain; sleep; congenital heart defect; surgery
MeSH Terms: conditions — Pain; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a randomized controlled crossover design. Research groups: 1. Swaddling group (control), 2. Swaddling combined with rocking and white noise feature in a multifunctional primary cradle group.
  In the crossover design, two groups were defined: Group A and Group B, where interventions were applied in different orders. Infants will be assigned to either group A or group B using a simple randomization method. The infant will be assigned to the control and experimental groups according to the order of initiation within the group to which the infant belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A (26 babies) :
  1. Monitoring in a multifunctional baby carrier for the first 3 hours (experiment)
  2. Monitoring in an open incubator for the next 3 hours (control)
  Interventions: Other: Multifunctional Baby Carrier
- Group B (Active Comparator): Group B (26 babies) :
  1. Monitoring in an open incubator for the next 3 hours (control)
  2. Monitoring in a multifunctional baby carrier for the first 3 hours (experiment)
  Interventions: Other: Multifunctional Baby Carrier

INTERVENTIONS:
Other: Multifunctional Baby Carrier — The study will be conducted using a randomized controlled crossover design. Infants will be assigned to either group A or group B using a simple randomization method. The infant will be assigned to the control and experimental groups according to the order of initiation within the group to which the infant belongs. Since the study is cross-over in design, infants in both groups (Group A and Group B) will be included in both the experimental group and the control group. Each baby will be monitored for a total of 6 hours.
  Group A (26 babies):
  1. Monitoring in a multifunctional main cradle during the first 3 hours (experiment)
  2. Monitoring in an open incubator wrapped for the second 3 hours (control)
  Group B (26 babies):
  1. Monitoring in an open incubator wrapped for the second 3 hours (control)
  2. Monitoring in a multifunctional main cradle during the first 3 hours (experiment)

SUMMARY:
The study aims to investigate the effect of using a multifunctional baby carrier with rocking, safe swaddling, and white noise features on physiological parameters, crying, and sleep status in infants aged 0-3 months who have undergone congenital heart surgery. It is planned to be conducted in a randomized controlled crossover design. Following congenital heart surgery, the use of sedative interventions in the high-stress environment of the intensive care unit has a significant effect on preserving the energy reserves necessary for the infant's growth and development. Using a sensitive and soothing mobile crib to assist in the postoperative care of infants who have undergone congenital heart surgery is a potential opportunity for the infant, nurse, and parent. The combined application of swaddling, sound, and movement reduces the baby's fussiness and has a calming effect on their physiological activation.

Infants who underwent heart surgery between 0-3 months and were followed up in a multi-purpose baby carrier (swaddling, white noise, and rocking) compared to infants in the follow-up experimental group, compared to infants in the control group who were only swaddled;

Hypothesis 1: The heart rate is lower. Hypothesis 2: Blood pressure is lower. Hypothesis 3: Oxygen saturation levels are higher. Hypothesis 4: Sleep durations are longer. Hypothesis 5: Pain scores are lower.

DETAILED DESCRIPTION:
This thesis study was designed to investigate the effect of using a multifunctional baby carrier with rocking, safe swaddling, and white noise features on physiological parameters, pain, crying, and sleep status in infants aged 0-3 months who underwent congenital heart surgery.

The sample size for the study, which is a 2x2 crossover design, was calculated using power analysis a large effect size and 80% power, resulting in a sample size of 52. Infants will be assigned to groups using simple randomization.

The dependent variables of the study are the infant's heart rate, blood pressure, oxygen saturation, sleep status, pain scale score, and crying duration. The independent variables are: the baby's gender, the baby's age, the postoperative day, the time spent at home with the parent, swaddling, white noise, and rocking.

Research groups: 1. Swaddling group (control), 2. Swaddling combined with rocking and white noise feature in a multifunctional primary cradle group.

In the crossover design, two groups were defined: Group A and Group B, where interventions were applied in different orders.

The data collection tools used in the study were the Infant Information Form, Infant Intervention Monitoring Form, Neonatal Pain, Agitation, and Sedation Scale (N PASS), Pediatric Sequential Organ Failure Assessment Score (pSOFA), Informed Consent Form-Parent Form, monitor , actigraph, stopwatch, decibel meter, swaddling cloth, and multi-functional baby carrier crib will be used as data collection tools in the study. Research data will be analyzed using the Statistical Package for Social Sciences (SPSS) program.

The safety of patients' vital sign data will be ensured through graphs. Pain assessment using the N-PASS scale will be evaluated by the same two observers, and inter-observer agreement will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Babies born at 38 weeks or later
* Babies aged 0 to 3 months after birth
* No illness other than congenital heart disease
* Who has undergone surgery for the first time due to congenital heart disease
* Whose clinical condition is stable (PSOFA score below 8 points)
* Infants with stable thermoregulation

Exclusion Criteria:

* Babies born before 38 weeks of pregnancy
* Babies older than 3 months
* The presence of other chromosomal or neurological disorders and syndromes in the infant
* Those who have undergone two or more surgeries due to congenital heart disease
* pSOFA score above 8 points

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Newborn Pain, Agitation and Sedation Scale (N PASS Scale) | 6 hours
  Term and preterm newborns are used for the purpose of evaluating postoperative pain/agitation and sedation. The total pain score ranges from 0 to +11. A high score indicates significant pain.
Sleep-Wake Status Measurement Device (Actigraphy) | 6 hours
  It is used to monitor babies' sleep-wake cycles.

SECONDARY OUTCOMES:
Pediatric Sequential Organ Failure Assessment Score (pSOFA) | 6 hours
  It is used to measure the severity of the disease and determine mortality. The lowest score is 0 and the highest score is 28 points. It is stated that mortality increases as the score increases. The Pediatric Sequential Organ Failure Assessment Score cutoff point distinguishing mortality is specified as 8 points. For this reason, infants with a pSOFA score below 8 points will be included in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Mutlu, Assc prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Health Sciences University Dr. Siyami Ersek Chest, Heart, and Vascular Surgery Education and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The consent forms stated that the confidentiality of the information would be protected and that it would be used only for the evaluation of the data in this study without identifying information.